CLINICAL TRIAL: NCT02747212
Title: Measuring the Electrical Properties of the Excised Malignant Tissues Obtained From Cancer Surgeries
Brief Title: Measuring the Electrical Properties of Malignant Tissues Ex Vivo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southern Medical University, China (Other)
Collaborators: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Sherman Xuegang Xin, Professor, Southern Medical University, China
Other Study IDs: SXXin-EPs-measurement-ex vivo
Record Dates: First submitted 2016-02-22; First posted 2016-04-21 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms
Keywords: electrical properties; malignant tissues; ex vivo
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: network analyzer — The dielectric properties of the tissues were measured using the open-ended coaxial line method. The measurement system consisted of a network analyzer (Model 4395A, Agilent Corp., Santa Clara, CA) associated with an S-parameter test set (Model 87511A, Agilent Corp., Santa Clara, CA). A semi-rigid coaxial line with a diameter of 3.58 mm was connected to the network analyzer system by using a Bayonet Neill-Concelman connector. The other tip of the coaxial line (probe) was placed on the flat bare surface of the tissue that placed on a measurements experiment platform.

SUMMARY:
Previously published studies have indicated that there exist difference in electrical properties (EPs), i.e., the conductivity and relative permittivity, between malignant and adjacent normal tissue, which will be useful in the early detection of cancers. While the EP informations of cancer tissues are not sufficient enough. The purpose of this study is to measure the electrical properties of the excised malignant tissues obtained from cancer surgeries.

DETAILED DESCRIPTION:
The measurements were conducted in the operating rooms of the hospital where the tissues were excised. Once the tissue was excised from the patient, the pathologist assisted the one of the engineers (already at the hospital) responsible to conduct the measurement. The specimen were designed to permit at least one measurement of malignant tissue and at least one measurement of normal tissue. Occasionally, the measurement of normal tissue was not possible if, for example, the normal tissue occupied a volume of small proportion for every excised specimen. The specimens for dielectric properties measurement were classified as normal or malignant by the pathologist based on his own expertise and decision criteria (visual inspection, anatomy) and the per-operative histological examination. The measurements were directly performed on the bulk specimen. The patient age, tissue temperature at the time of measurement and time between excision and measurement for each sample were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer Disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who are diagnosed with cancer disease and about to have an operation to excise the cancer tissues
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Conductivity of Malignant Tissues Measured Ex Vivo | one year
Relative Permittivity of Malignant Tissues Measured Ex Vivo | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sherman X Xin, professor, Principal Investigator — School of Biomedical Engineering,Southern Medical University
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Athey T W, Stuchly M A and Stuchly S S. Measurement of radio frequency permittivity of biological tissues with an open-ended coaxial line: Part I. Microwave Theory and Techniques, IEEE Transactions on IEEE Trans 30(1): 82-86, 1982.
- [Background] Bobowski Jake S, Johnson Thomas. Permittivity measurements of biological samples by an open-ended coaxial line. Progress In Electromagnetics Research B 40: 159-183, 2012.
- [Background] Surowiec AJ, Stuchly SS, Barr JB, Swarup A. Dielectric properties of breast carcinoma and the surrounding tissues. IEEE Trans Biomed Eng. 1988 Apr;35(4):257-63. doi: 10.1109/10.1374. No abstract available. PMID 2834285
- [Background] Smith SR, Foster KR, Wolf GL. Dielectric properties of VX-2 carcinoma versus normal liver tissue. IEEE Trans Biomed Eng. 1986 May;33(5):522-4. doi: 10.1109/TBME.1986.325740. No abstract available. PMID 3710509
- [Background] Mehta P, Chand K, Narayanswamy D, Beetner D G, Zoughi R and Stoecker W V. Microwave reflectometry as a novel diagnostic tool for detection of skin cancers IEEE Trans. Instrum. Meas. 55: 1309-16, 2006
- See also: An Internet resource for the calculation of the dielectric properties of body tissues in the frequency range 10 Hz - 100 GHz Based on data published by C.Gabriel et al. in 1996. — http://niremf.ifac.cnr.it/tissprop/